CLINICAL TRIAL: NCT04553094
Title: Evaluation of the Effects of Personalized Training at Home Combining Endurance and Resistance in Patients Suffering From Marfan Syndrome
Brief Title: Effects of Personalized Training at Home Combining Endurance and Resistance in Patients Suffering From Marfan Syndrome
Acronym: MARF'HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-01
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Marfan Syndrome
Keywords: Physical training
MeSH Terms: conditions — Marfan Syndrome | interventions — Endurance Training

STUDY DESIGN:
Intervention Model Description: 3 groups of physical training intervention compared with control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (No Intervention): No physical training
- Group 2 (Experimental): Endurance training
  Interventions: Other: Endurance training
- Group 3 (Experimental): Muscle building training
  Interventions: Other: Muscle building training
- Group 4 (Experimental): Training combining endurance + muscle building
  Interventions: Other: Endurance training; Other: Muscle building training

INTERVENTIONS:
Other: Endurance training — Aerobic circuit training
  Arms: Group 2; Group 4
Other: Muscle building training — Muscle strengthening circuit training
  Arms: Group 3; Group 4

SUMMARY:
Marfan syndrome (MS) is an autosomal dominant genetic disorder caused by a mutation in the fibrillin-1 gene (FBN1) encoding the protein fibrillin-1. Fibrillin is the main component of microfibrils, elements found in all of the body's tissues, and this pathology is characterized by the multitude of its clinical manifestations. These patients may develop aneurysms in the aortic root and one of the main factors of morbidity in patients with MS is aortic dissection. Prevention mainly involves preventive aortic surgery. However, the repercussions are global and can affect the functioning of other tissues such as skeletal muscle tissue, bone tissue, lung tissue and the eyes. The association of skeletal (scoliosis, hyperlaxity), muscular and ocular disorders is clearly associated with an impairment in the quality of life. These disorders are associated with pain and disability which affect professional activity, leisure and family life.

Physical activity could represent a relevant alternative for these patients. A recent animal study suggests that moderate training is beneficial.

DETAILED DESCRIPTION:
The main objective is to show that the quality of life of patients with Marfan syndrome can be improved by personalized training at home. The goal is to be able to offer new non-drug management based on physical activity to these patients.

Improved quality of life; Improvement of muscle strength by a muscle strengthening protocol; Improvement of cardiovascular function parameters. Regular coaching throughout the study.

1. / Assessment of muscular capacities
2. / Assessment of cardiovascular and respiratory capacities
3. / Response to psychometric questionnaires
4. / Participation in a training circuit (training protocol)

ELIGIBILITY:
Inclusion Criteria:

* patient with Marfan syndrome and followed up at Bichat Claude Bernard hospital, Paris. Marfan syndrome should be diagnosed according to the Ghent nosology revised in 2010
* Patient taking protective treatment for the aorta (beta blocker, calcium channel blocker, ACE inhibitor, angiotensin II receptor antagonist).
* Valid patient, able to return to consultation and carry out functional assessments and personalized physical training at home.
* Patients operated prophylactically on the ascending aorta may be included at a distance > 6 months from their surgery.

Exclusion Criteria:

* Myocardial pathology other than Marfan syndrome.
* Thoracic aorta dissection.
* Aortic diameter > 45 millimeters.
* Uncontrolled high blood pressure at rest (systolic blood pressure > 140 Millimeter of mercury and diastolic blood pressure > 90 Millimeter of mercury)
* Increase in systolic blood pressure > 160 Millimeter of mercury during exercise.
* Pregnancy at the time of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Quality of life assessment: questionnaire | 3 months
  Assessed with Medical Outcome Study Short Form 36 questionnaire, a scale scored on a 0 to 100 range so that the lowest is the worth condition and highest is the best condition.

SECONDARY OUTCOMES:
Pain assessment: Fibromyalgia Rapid Screening Tool | 3 months
  Assessed with Fibromyalgia Rapid Screening Tool
Self-perception assessment | 3 months
  Assessed with Physical Self Inventory questionnaire, a scale scoring 25 items rated on a 6-point scale ranging from 1 (Not at all) to 6 (Entirely) and assessing 6 dimensions (global self-worth (10-50), physical self-worth (10-50), physical condition (10-50), sport competence (10-40), physical attractiveness (10-30), and physical strength (10-30)) of the physical self-conception.
Aortic diameter | 3 months
  Evolution of the aortic diameter (in millimeter) in echocardiography, safety cardiovascular parameters
Blood pressure | 3 months
  Evolution of the systolic and diastolic blood pressures (in Millimeter of mercury) during exercise, monitoring of physiological parameters
Heart rate | 3 months
  Evolution of heart rate (Beats per minute) during exercise, monitoring of physiological parameters
oxygen consumption | 3 months
  Evolution of oxygen consumption (in liter) during exercise, monitoring of physiological parameters
Maximal voluntary contraction | 3 months
  Evolution of maximal voluntary contraction (in Newtons) during exercise, monitoring of physiological parameters
Left Ventricular Ejection Fraction (LVEF) | 3 months
  Evolution of Left Ventricular Ejection Fraction (in percentage) at rest, monitoring of cardiovascular parameters.
Global longitudinal strain (GLS) | 3 months
  Evolution of GLS (in percentage) at rest, monitoring of cardiovascular parameters

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume JONDEAU, MD, Principal Investigator — Groupe Hospitalier Bichat - Claude Bernard
Locations (1):
- Groupe Hospitalier Bichat - Claude Bernard, Paris, France

REFERENCES:
- [Derived] Jouini S, Milleron O, Eliahou L, Jondeau G, Vitiello D. Online Personal Training in Patients With Marfan Syndrome: A Randomized Controlled Study of Its Impact on Quality of Life and Physical Capacity. J Am Heart Assoc. 2024 Oct;13(19):e033024. doi: 10.1161/JAHA.123.033024. Epub 2024 Sep 18. PMID 39291498